CLINICAL TRIAL: NCT00300690
Title: Choice of Material for Above-Knee Femoro-Popliteal Bypass Prosthetic Graft. Multicenter Randomized Study of an Impregnated Knitted Polyester Prosthesis Vs. PTFE (Uni-Graft Vs Gore-Tex).
Brief Title: Choice of Material for Above-Knee Femoro-Popliteal Bypass Prosthetic Graft (PopUp)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C124
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2006-03-09 (Estimated); Status verified 2006-03

CONDITIONS: Intermittent Claudication; Critical Limb Ischemia
Keywords: Lower extremity bypass surgery; femoro-popliteal bypass; Dacron material; PTFE material
MeSH Terms: conditions — Intermittent Claudication; Chronic Limb-Threatening Ischemia

INTERVENTIONS:
Device: 6 mm Uni-graft® (B-Braun)
Device: 6 mm Gore-Tex® (WL Gore)

SUMMARY:
This trial was designed to challenge the wide held view that polytetrafluoroethylene (PTFE) performs better than Dacron for above knee femoropopliteal bypass.

DETAILED DESCRIPTION:
Objective: To investigate whether patency rates of 6 mm gelatine coated, knitted, double velour polyester prostheses are equal to the 6 mm thinwalled ePTFE prostheses as above-knee femoro-popliteal bypass graft

ELIGIBILITY:
Inclusion Criteria:

* All patients who require revascularisation of the lower extremity suitable for above-knee femoro-popliteal bypass surgery.

Exclusion Criteria:

* pregnancy
* No consent to participate in the study
* Previous enrollment in the study
* follow-up is not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1993-10; Study Completion 1999-01

PRIMARY OUTCOMES:
Primary uncorrected graft patency after 2 years

SECONDARY OUTCOMES:
- Secondary graft patency after two years
- Limb survival after two years
- Complication rate perioperatively

CONTACTS AND LOCATIONS:
Overall Officials: Torben V Schroeder, Professor, Principal Investigator — Rigshospitalet, Denmark